CLINICAL TRIAL: NCT01767493
Title: An Open-label, Non-randomized Study to Evaluate the Feasibility of [18F]Florbetapir Positron Emission Tomography (PET) for Assessment of Demyelination in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Study to Evaluate the Feasibility of [18F]Florbetapir PET for Assessment in MS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Florbetapir MS 01
Record Dates: First submitted 2012-12-13; First posted 2013-01-14 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]Florbetapir PET imaging (Experimental): [18F]Florbetapir and PET imaging
  Interventions: Drug: [18F]Florbetapir PET imaging

INTERVENTIONS:
Drug: [18F]Florbetapir PET imaging — [18F]Florbetapir and PET imaging
  Other Names: Amyvid

SUMMARY:
The purpose of this study is to evaluate the feasibility of [18F]Florbetapir positron emission tomography (PET) for assessment of demyelination in the patients with relapsing remitting multiple sclerosis.

DETAILED DESCRIPTION:
The underlying goal of this study is to assess the feasibility of [18F]Florbetapir as an imaging tool to detect demyelination in the brain of MS research participants and compare to similarly aged healthy subjects.

ELIGIBILITY:
Eligibility criteria (for all subjects):

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local subject privacy regulations
* Willingness to comply with study procedures
* Willingness to provide written informed consent
* Age greater than or equal to 18 and less than or equal to 60 years old at the time of the informed consent
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception until PET testing is completed
* For females, must be of non-childbearing potential or have a negative urine and blood pregnancy test on the day of [18F]Florbetapir PET injection

Inclusion Criteria (Healthy Volunteers):

* No history of or signs of acute or chronic neurological or psychiatric illness based on evaluation by a research physician.

Inclusion Criteria (MS Subjects):

* Have a diagnosis of relapsing remitting MS according to the 2010 MacDonald Criteria
* Have at least 10 demyelinating lesion on brain MRI with the following characteristics:
* Hypointense on T2 weighted images with FLAIR

Exclusion Criteria (for all subjects):

* The subject has clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological (other than RRMS), immunodeficiency, pulmonary, or other disorder or disease.
* Women who are pregnant or actively breastfeeding
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery)
* The subject has participated in another clinical study within the previous 30 days
* Renal impairment with a creatine clearance <80mL/minute at screening (creatine clearance estimated by Cockcroft-Gault equation)
* The subject is scheduled to have a major surgery or procedure during the time of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- See also: Institute for Neurodegenerative Disorders — http://www.indd.org

RESULTS

PARTICIPANT FLOW:
Groups:
- [18F]Florbetapir Imaging: [18F]Florbetapir and PET imaging
Period: Overall Study
Arm/Group | [18F]Florbetapir Imaging
Started | 19
Completed | 16
Not Completed | 3
Not completed — screen failures | 3

BASELINE CHARACTERISTICS:
Arm/Group | [18F]Florbetapir PET Imaging
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Lesions Detected by [18F]Florbetapir PET
Description: This study demonstrates the feasibility of[18F]Florbetapir PET for identifying demyelinating lesions in relapsing-remitting MS patients. It was expected that lesion size played a factor in identifying white matter lesions with those smaller than 5 mm less evident on PET. Using spherical volumes of interest the extent of reduction in the white matter uptake can be reliably quantified. This requires careful attention to techniques for sampling in both the lesions and white matter control regions for the subject.
Time Frame: 1 year
Measure: Number; unit: Lesions
Arm/Group | [18F]Florbetapir PET Imaging
Number analyzed (Participants) | 19
Lesions | 194

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 year.
Description: There were three adverse events and all three were considered to be unrelated to the imaging or other study procedures.
Arm/Group | [18F]Florbetapir PET Imaging
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 2/19
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [18F]Florbetapir PET Imaging (N=19)
Wrist Pain (Injury, poisoning and procedural complications) | 1 (1) — The pain was deemed unrelated to imaging or other study procedures. The pain was mild and not limiting.
Chest Wall Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — The adverse event was mild. The adverse event was deemed unrelated to imaging or other study procedures. The AE has been resolved.
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 (1) — The adverse event was mild and deemed unrelated to imaging or other study procedures. The AE has been resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes